CLINICAL TRIAL: NCT05321875
Title: Early Treatment With Candesartan vs Placebo in Asymptomatic Genetic Carriers of Dilated Cardiomyopathy (EARLY-GENE Trial)"
Brief Title: Early Treatment With Candesartan vs Placebo in Genetic Carriers of Dilated Cardiomyopathy (EARLY-GENE Trial)
Acronym: EARLY-GENE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cristina Avendaño Solá (Other)
Responsible Party: Sponsor-Investigator, Cristina Avendaño Solá, Head of Clinical Pharmacology Department, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EARLY-GENE; 2021-004577-30 (EudraCT Number)
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Cardiomyopathy, Dilated
Keywords: Dilated Cardiomyopathy; Genetic Mutation Carrier; Randomized Clinical Trial; Genetic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — candesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical placebo tablets manufactured by the same Manufacturer of active marketed Candesartan (KERN PHARMA). Double-blind labelling specific for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Candesartan (Experimental): Candesartan, 16 mg oral tablets. Target dose 32 mg or maximum tolerated dose after dose escalation from 16 mg
  Interventions: Drug: Candesartan
- Placebo (Placebo Comparator): Matching placebo. Target dose 2 tablets or maximum tolerated dose after dose escalation from 1 tablet
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Candesartan — 3 years treatment with candesartan target dose: 32 mg or maximum tolerated dose after dose escalation from 16 mg

SUMMARY:
Prospective, multicenter, randomized, placebo-controlled, double-blind clinical trial to evaluate safety and efficacy of candesartan in the prevention of the development of Dilated Cardiomyopathy (DCM) in genetic carriers of a DCM-causing variant without disease expression (asymptomatic)

DETAILED DESCRIPTION:
Prospective, multicenter, randomized, placebo-controlled, double-blind clinical trial to evaluate safety and efficacy of early administration of candesartan in the prevention of the development of Dilated Cardiomyopathy (DCM) in genetic carriers of a DCM-causing variant without disease expression (asymptomatic).

Randomization will be 1:1 and patients are allocated to candesartan or matching placebo.

Patients will be followed for a 3 years period and efficacy will be demonstrated if candesartan (compared to placebo) prevents either a significant Left ventricular ejection fraction (LVEF) decline of ≥10%, or a ventricular dilatation (left ventricular end-diastolic volume, LVEDV) increase of ≥10% within a 3-years period of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-64 (both included), both sexes
* Carrier of a pathogenic or likely pathogenic DCM genetic variant1 according to modified American College of Medical Genetics (ACMG) criteria.
* Baseline LVEF ≥ 50% measured by MRI1 and evaluated by the eligibility study committee. Carriers with myocardial fibrosis, detected by late gadolinium enhancement in magnetic resonance imaging, are valid.
* Baseline creatinine ≤1.3 mg/dL, potassium ≤ 5.3 mEq/L and an estimated Glomerular Filtration Rate (eGFR)≥ 60 ml/min/1.73 m2 calculated by CKD-EPI formula.
* Able to understand and accept the study constraints and to provide informed consent.

Exclusion Criteria:

* Hypotension (systolic arterial pressure <100 mmHg (measured following a standardized methodology).
* Prior ventricular dysfunction (LVEF ≤ 50% at any time prior to study inclusion)
* Candidates who are expected or highly likely to receive an implantable cardioverter defibrillator (ICD) in the following 12 months after inclusion in the trial
* Preexisting hypertension requiring pharmacological treatment.
* Uncontrolled arterial hypertension (i.e., repeatedly systolic arterial pressure > 140 mmHg).
* Carriers of TTN-truncating variants (TTNtv) who are < 35 years old.
* Known clinically significant coronary artery disease (e.g., ≥70% stenosis in any epicardial artery or ≥50% of left main coronary artery), valvular disease (≥ moderate in severity) or ventricular arrhythmias.
* Ongoing treatment with ACEI, ARB, ARNI or MRA.
* Prior intolerance to ACE inhibitors or ARB.
* Presence of any contraindications to receive candesartan treatment, including severe liver failure and/or cholestasis
* Known bilateral renal artery stenosis.
* Uncontrolled concomitant severe disease (e.g., with expected survival inferior to the duration of the study follow-up)
* Participation in any other clinical trial using an investigational medicinal product or device in the 30 days previous to the inclusion in the study.
* Current pregnancy, breastfeeding or women of childbearing age who are not willing to practice an adequate birth control during the entire duration of the study (a negative pregnancy test result must be confirmed at the time of enrolment)*.
* Drug or alcohol abuse (current).
* Inability to comply with study procedures and treatments.
* Carriers of MRI incompatible internal devices (ICD, pacemakers, aneurysm clips, etc.), with known intolerance to MRI studies or presenting any contraindications to perform cardiac MRI studies.
* Any circumstances that in the investigator's opinion compromise the participant's ability to participate in the clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants that progress to either a LVEF or LVEDV deterioration of ≥10% with respect to the baseline value at the end of follow-up as measured by MRI | 3 years

SECONDARY OUTCOMES:
Proportion of participants that progress to a LVEF deterioration of ≥10% compared to baseline value at the end of follow-up as measured by MRI. | 3 years
Proportion of participants that progress to a LVEDV deterioration of ≥10% compared to baseline value at the end of follow-up as measured by MRI. | 3 years
Changes in LVEF measured by MRI (vs baseline) | 3 years
Changes in LVEDV measured by MRI (vs baseline) | 3 years
Proportion of individuals who develop DCM (LVEF<50%). | 3 years
Proportion of participants in each treatment group developing Serious Adverse Events (SAEs), Grade 3-4 adverse events (AEs), Adverse Reactions, or AEs of Special Interest (AESIs). | 3 years
Proportion of treatment discontinuations in the candesartan and placebo groups. | 3 years

OTHER OUTCOMES:
Proportion of participants developing new cardiac fibrosis and its extent measured by MRI in the candesartan and placebo groups. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pablo García-Pavía, MD, PhD, Study Chair — Hospital Universitario Puerta de Hierro Majadahonda
Locations (1):
- Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under agreement, individual or aggregated patient data could be shared with other scientific groups for new scientific projects. Data can be shared only for scientific purposes and in full compliance with Personal Data Protection requirements in the EU
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study scientific publication
Access Criteria: Under request to Study Chair